CLINICAL TRIAL: NCT01964001
Title: The Effects of Vitamin B-6 and Coenzyme Q10 Status on Oxidative Stress, Antioxidant Capacities, and Inflammatory Responses in Patients With Liver Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CF13197
Record Dates: First submitted 2013-10-10; First posted 2013-10-17 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Hepatocellular Carcinoma.
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Vitamin B 6; coenzyme Q10

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): starch
  Interventions: Other: Placebo
- Dietary supplements (Experimental): Vitamin B-6/Coenzyme Q10/vitamin B6+Coenzyme Q10
  Interventions: Dietary Supplement: Vitamin B-6; Dietary Supplement: Coenzyme Q10; Dietary Supplement: Vitamin B-6+Coenzyme Q10

INTERVENTIONS:
Dietary Supplement: Vitamin B-6 — Vitamin B-6 50 mg/d
  Arms: Dietary supplements
Dietary Supplement: Coenzyme Q10 — Coenzyme Q10 300 mg
  Arms: Dietary supplements
Dietary Supplement: Vitamin B-6+Coenzyme Q10 — Vitamin B-6 (50 mg/d) and Coenzyme Q10 (300 mg/d)
  Arms: Dietary supplements
Other: Placebo — starch
  Arms: Placebo

SUMMARY:
Carcinoma is the leading cause of worldwide. Hepatocellular carcinoma (HCC) is the second cause of cancer mortality in Taiwan. Vitamin B-6 and coenzyme Q10 has been recognized as antioxidants and anti-inflammatory nutrients in recent clinical studies. The purposes of this study are going to investigate the relation of vitamin B-6 and coenzyme Q10 with the indicators of oxidative stress, antioxidant enzymes activities and the inflammatory markers in patients with stage 1 and stage 2 HCC. The study is designed as an intervention study. The investigators will recruit HCC patients with stage 1 and stage 2 (n = 150) who are identified by liver biopsy. HCC subjects are randomly assign to placebo, vitamin B-6 (50 mg/d), coenzyme Q10 (300 mg/d), and vitamin B-6 plus coenzyme Q10 supplements groups. Intervention is going to administration for three months. The concentrations of vitamin B-6, coenzyme Q10, oxidative stress indicators, antioxidant enzymes activities, antioxidant vitamins (vitamin A and E), and inflammatory markers are going to be analyzed. The results would provide more information nutrients for clinical physicians and dietitians for considering suggesting patients with HCC using vitamin B-6 or coenzyme Q10 supplementation to improve their clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

- The HCC patients with stage 1 and stage 2 (n = 150) who are identified by liver biopsy.

Exclusion Criteria:

* age < 20 years old.
* The patients who had heart, renal, gestational, diabetes, or other metabolic diseases.
* Under the medications which may interfere the vitamin B-6 or coenzyme Q10 concentrations, such as phenobarbital, phenytoin, cycloserine, pyrazinamide, isoniazid, (thio)semicarbazide, hydramitrazine, phenelzine, carbidopa, levodopa, hydralazine, steroids, penicillamine, ,Statin, or Warfarin.
* The women who are during pregnancy or Lactation.
* The women who are taking the oral contraceptives.
* The subjects who are taking the dietary supplements, such as vitamin B-6, coenzyme Q10, or other antioxidant vitamins.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Antioxidant capacity | 12 weeks
  This study are going to measure the indicators of antioxidant capacity including Vitamin B-6, coenzyme Q10, vitamin A and E, lipid peroxidation markers (malondialdehyde), and antioxidant enzymes activities (catalase, glutathione peroxidase and superoxide dismutase).

SECONDARY OUTCOMES:
Inflammation markers | 12 weeks
  This study are going to measure the inflammation markers including C-reactive protein, Tumor necrosis factor-alfa, Interleukin-1 beta, Interleukin-6,adiponectin, homocysteine, S-adenosyl-methionine, and S-adenosyl-homocysteine.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Verterans General Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Liu HT, Huang YC, Cheng SB, Huang YT, Lin PT. Effects of coenzyme Q10 supplementation on antioxidant capacity and inflammation in hepatocellular carcinoma patients after surgery: a randomized, placebo-controlled trial. Nutr J. 2016 Oct 6;15(1):85. doi: 10.1186/s12937-016-0205-6. PMID 27716246
- [Derived] Cheng SB, Lin PT, Liu HT, Peng YS, Huang SC, Huang YC. Vitamin B-6 Supplementation Could Mediate Antioxidant Capacity by Reducing Plasma Homocysteine Concentration in Patients with Hepatocellular Carcinoma after Tumor Resection. Biomed Res Int. 2016;2016:7658981. doi: 10.1155/2016/7658981. Epub 2016 Mar 9. PMID 27051670